CLINICAL TRIAL: NCT03858933
Title: Train Your Brain: A Neurofeedback Intervention for Individuals With Post-Traumatic Stress Disorder
Brief Title: Train Your Brain: Neurofeedback Intervention for PTSD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Regulations
Sponsor: University of Southern California (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Jeremy Goldbach, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UP-16-00399-AM011
Record Dates: First submitted 2018-11-16; First posted 2019-03-01 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: PTSD; Post-Traumatic Stress Disorder; Acute Stress Syndrome; Emotion Regulation; Depression; Anxiety; Sexual Assault; Combat PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Emotional Regulation; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The eBrainFit Platform is set to randomize each entered Subject Identification Number into either the alpha/theta or limbic modulation treatment arms. Neither the participant nor researcher will know the arm, to which the participant has been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Limbic Modulation Index Neurofeedback (Experimental): This arm of the study will undergo a novel neurofeedback treatment, targeting downregulation of deep limbic structures, specifically the amygdalae.
  Participants in this arm will complete 15 neurofeedback sessions.
  Interventions: Device: eBrainFit Platform
- Alpha/Theta Neurofeedback (Active Comparator): This arm of the study will undergo a proven PTSD neurofeedback treatment, alpha/theta regulation, during which participants will try various mental strategies to increase the presence of theta waves.
  Participants in this arm will complete 15 neurofeedback sessions.
  Interventions: Device: eBrainFit Platform

INTERVENTIONS:
Device: eBrainFit Platform — Alpha/Theta regulation with eyes open
  Arms: Alpha/Theta Neurofeedback
Device: eBrainFit Platform — Amygdala regulation with eyes open
  Arms: Limbic Modulation Index Neurofeedback

SUMMARY:
The investigator's aim is to evaluate the efficacy of two types of neurofeedback treatments for PTSD symptoms reduction. Half of the participants will receive the current standard for PTSD neurofeedback care undergoing alpha/theta neurofeedback regulation. The other half will receive the newly developed limbic modulation index neurofeedback.

DETAILED DESCRIPTION:
Traumatic stress is commonly resistant to existing therapeutics, possibly due to high treatment dropout rates along with a failure to target the relevant underlying neural mechanisms. Neuromodulation of deep limbic areas such as the amygdala may play a critical role in the effective recovery from traumatic stress. Human studies have shown the importance of such modulation during the encoding of traumatic stimuli, showing greater amygdala activation for subsequently remembered traumatic stimuli. In addition, a prospective study among previously healthy soldiers showed that hyper-activation of the amygdala prior to military traumatic exposure corresponded with more severe post-traumatic symptoms following exposure.

Together these finding points to the amygdala as a plausible neuromodulation target for preventive or early interventions of post-traumatic disturbances. Local neuromodulation of the amygdala could improve treatment specificity and the overall intervention outcome.

The main goal of the suggested research is to further develop and implement a non-invasive, portable and cost-effective brain-imaging tool that will provide individual on-line guidance for amygdala modulation. This closed-loop brain training will enhance individual resilience to and coping with potentially traumatic stress as well as alleviate consequential psychopathologies.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of PTSD
* PTSD symptoms within the last 30 days

Exclusion Criteria:

* Any active psychosis or suicidal intent
* A severe traumatic brain injury (one in which consciousness was lost for greater than 6 hours)
* Any of the following neurological disorders: Parkinson's, Alzheimer's, Brain Tumor, or Brain Lesion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline PTSD severity using the Clinician Administered PTSD Scale for Diagnostic and Statistical Manual of Mental Disorders-5 | administered at Initial Appointment (Week 0) and one week after the 15th neurofeedback session (approximately Week 22).
  The five-point CAPS-5 symptom severity rating scale is used for all symptoms. Rating scale anchors should be interpreted and used as follows:
  0 Absent The respondent denied the problem or the respondent's report doesn't fit the DSM-5 symptom criterion.
  1. Mild / subthreshold:
  2. Moderate / threshold:
  3. Severe / markedly elevated:
  4. Extreme / incapacitating:
  CAPS-5 total symptom severity score is calculated by summing severity scores for items 1-20.
  CAPS-5 symptom cluster severity scores are calculated by summing the individual item severity scores for symptoms contained in a given DSM-5 cluster.

SECONDARY OUTCOMES:
Emotion Regulation Questionnaire | administered at Initial Appointment (Week 0), Start of Neurofeedback (Week 7) and one week after the 15th neurofeedback session (approximately Week 22)
  A 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal and (2) Expressive Suppression. Respondents answer each item on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree).
  Items 1, 3, 5, 7, 8, 10 make up the Cognitive Reappraisal facet. Items 2, 4, 6, 9 make up the Expressive Suppression facet. Scoring is kept continuous. Each facet's scoring is kept separate.
Beck Depression Inventory | administered at Initial Appointment (Week 0), Start of Neurofeedback (Week 7) and one week after the 15th neurofeedback session (approximately Week 22)
  Quantifies depressive symptoms using a 21-item measure.
  Depression severity is calculated by summing the score responses, with higher values indicating more severe symptom expression.
Beck Anxiety Inventory | administered at Initial Appointment (Week 0), Start of Neurofeedback (Week 7) and one week after the 15th neurofeedback session (approximately Week 22)
  Quantifies anxious symptoms using a 21-item measure
  Anxiety severity is calculated by summing the score responses, with higher values indicating more severe symptom expression.
PTSD Checklist for DSM-5 | administered at Initial Appointment (Week 0), Start of Neurofeedback (Week 7) and one week after the 15th neurofeedback session (approximately Week 22)
  Quantifies PTSD symptoms using a 20-item measure
  PTSD severity is calculated by summing the score responses, with higher values indicating more severe symptom expression.
Sleep Duration | administered at Initial Appointment (Week 0), Start of Neurofeedback (Week 7) and one week after the 15th neurofeedback session (approximately Week 22)
  Captured using a Fitbit Physical Activity Tracking Device
  The device will report the participant's sleep duration (output in minutes) for each night the device is worn.
Emotional Stroop Task | administered at Initial Appointment (Week 0), Start of Neurofeedback (Week 7) and one week after the 15th neurofeedback session (approximately Week 22)
  Behavioral metric of conflict adaptation.
  Emotion regulation will be assessed using a well-established emotional conflict paradigm that arises from an incompatibility between the task-relevant and task-irrelevant emotional dimensions of a stimulus and allows for the tracking of emotion regulation from trial to trial. In this task there is less conflict, indexed by faster reaction times for incongruent trials, than if they are preceded by a congruent trial. This difference in reaction times between low conflict resolution and high conflict resolution trials serves as a behavioral metric of conflict adaptation. A negative adaptation score reflects activation of a regulatory mechanism that leads to improved emotional conflict resolution.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Goldbach, PhD, Principal Investigator — Faculty Professor
Locations (1):
- University Of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Online Eligibility Survey — https://uscsocialwork.qualtrics.com/jfe/form/SV_2b397uP7BK75yUR

DOCUMENTS (1):
  • Informed Consent Form (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT03858933/ICF_000.pdf